CLINICAL TRIAL: NCT04478266
Title: A Randomized, Multicenter, Double-blind Phase 3 Study of Amcenestrant (SAR439859) Plus Palbociclib Versus Letrozole Plus Palbociclib for the Treatment of Patients With ER (+), HER2 (-) Breast Cancer Who Have Not Received Prior Systemic Anti-cancer Treatment for Advanced Disease
Brief Title: Amcenestrant (SAR439859) Plus Palbociclib as First Line Therapy for Patients With ER (+) HER2(-) Advanced Breast Cancer
Acronym: AMEERA-5
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated based on the review by an independent data monitoring committee of the prespecified interim analysis of the Phase 3 AMEERA-5 efficacy data. No new safety signals were observed.
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC15935; 2020-001824-33 (EudraCT Number); U1111-1233-0486 (Other: UTN)
Record Dates: First submitted 2020-07-10; First posted 2020-07-20 (Actual); Results first posted 2023-07-06 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; Letrozole; Goserelin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Letrozole + Palbociclib (Active Comparator): Participants received letrozole 2.5 milligrams (mg) capsule along with amcenestrant-matching placebo once daily, continuously and palbociclib 125 mg orally (PO), once daily (QD) from Day 1 to Day 21 of each 28-day treatment cycle until disease progression, death or study cut-off date, whichever comes first (maximum exposure: 112 weeks). Goserelin once every 4 weeks in pre/peri menopausal women and men.
  Interventions: Drug: Amcenestrant-matching placebo; Drug: Palbociclib; Drug: Letrozole; Drug: Goserelin
- Amcenestrant + Palbociclib (Experimental): Participants received amcenestrant 200 mg tablet along with letrozole-matching placebo once daily, continuously and palbociclib 125 mg PO, QD from Day 1 to Day 21 of each 28-day treatment cycle until disease progression, death, or study cut-off date, whichever comes first (maximum exposure: 109 weeks). Goserelin once every 4 weeks in pre/peri menopausal women and men.
  Interventions: Drug: SAR439859; Drug: Palbociclib; Drug: Goserelin; Drug: Letrozole-matching placebo

INTERVENTIONS:
Drug: Amcenestrant-matching placebo — Pharmaceutical form: Tablets Route of Administration: Oral
  Arms: Letrozole + Palbociclib
Drug: SAR439859 — Pharmaceutical form: Tablets Route of Administration: Oral
  Other Names: Amcenestrant
  Arms: Amcenestrant + Palbociclib
Drug: Palbociclib — Pharmaceutical form: Capsules/Tablets Route of Administration: Oral
  Other Names: Ibrance
Drug: Letrozole — Pharmaceutical form: Capsules Route of Administration: Orally
  Arms: Letrozole + Palbociclib
Drug: Goserelin — Pharmaceutical form: Depot Injection Route of Administration: Subcutaneous
Drug: Letrozole-matching placebo — Pharmaceutical form: Capsules Route of Administration: Orally
  Arms: Amcenestrant + Palbociclib

SUMMARY:
Primary Objective:

To determine whether Amcenestrant (SAR439859) in combination with palbociclib improves progression free survival (PFS) when compared with letrozole in combination with palbociclib in participants with estrogen receptor positive (ER+), human epidermal growth factor receptor 2 negative (HER2-) advanced breast cancer who have not received any prior systemic anticancer therapies for advanced disease.

Secondary Objective:

* To compare the overall survival in both treatment arms.
* To evaluate the objective response rate in both treatment arms.
* To evaluate the duration of response in both treatment arms.
* To evaluate the clinical benefit rate in both treatment arms.
* To evaluate progression-free survival on next line of therapy.
* To evaluate the pharmacokinetics of amcenestrant, and palbociclib.
* To evaluate health-related quality of life in both treatment arms.
* To evaluate the time to first chemotherapy in both treatment arms.
* To evaluate safety in both treatment arms.

DETAILED DESCRIPTION:
Study duration per participant was approximately 59 months, which includes a 33- month treatment period.

ELIGIBILITY:
Inclusion criteria :

* Adult participants with loco-regional recurrent or metastatic disease not amenable to curative treatment.
* Confirmed diagnosis of ER+/HER2- breast cancer.
* No prior systemic treatment for loco-regional recurrent or metastatic disease.
* Measurable disease evaluable per Response Evaluation Criterion in Solid Tumors (RECIST) v.1.1 or non-measurable bone-only disease.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Participants should be willing to provide tumor tissue.
* Capable of giving informed consent.

Exclusion criteria:

* Known active brain metastases.
* Prior neo (adjuvant) treatment with any selective estrogen receptor degrader (SERD).
* Inadequate organ and marrow function.
* Disease recurrence while on, or within 12 months of completion of (neo)adjuvant endocrine therapy.
* Pregnant, breastfeeding, or woman of childbearing potential unwilling to use recommended contraception methods.
* Male participants who disagree to follow contraception.
* Participants with advanced, symptomatic visceral spread, that are at risk of life-threatening complications in the short term.
* Participants with significant concomitant illness.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1068 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2023-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (249):
- United States (45):
  - Investigational Site Number :8400075, Daphne, Alabama
  - Investigational Site Number :8400083, Glendale, Arizona
  - Investigational Site Number :8400066, Tucson, Arizona
  - Investigational Site Number :8400038, Fullerton, California
  - Investigational Site Number :8400056, Los Alamitos, California
  - Investigational Site Number :8400029, Santa Monica, California
  - Investigational Site Number :8400025, Denver, Colorado
  - Investigational Site Number :8400059, Lakeland, Florida
  - Investigational Site Number :8400053, Orlando, Florida
  - Investigational Site Number :8400081, Palm Bay, Florida
  - Investigational Site Number :8400055, Athens, Georgia
  - Investigational Site Number :8400016, Atlanta, Georgia
  - Investigational Site Number :8400034, Savannah, Georgia
  - Investigational Site Number :8400035, Thomasville, Georgia
  - Investigational Site Number :8400039, Chicago, Illinois
  - Investigational Site Number :8400008, Fort Wayne, Indiana
  - Investigational Site Number :8400006, Iowa City, Iowa
  - Investigational Site Number :8400013, Westwood, Kansas
  - Investigational Site Number :8400028, Scarborough, Maine
  - Investigational Site Number :8400017, Boston, Massachusetts
  - Investigational Site Number :8400076, Danvers, Massachusetts
  - Investigational Site Number :8400077, Newton, Massachusetts
  - Investigational Site Number :8400002, Ann Arbor, Michigan
  - Investigational Site Number :8400005, Kansas City, Missouri
  - Investigational Site Number :8400004, St Louis, Missouri
  - Investigational Site Number :8400058, Las Vegas, Nevada
  - Investigational Site Number :8400015, New Brunswick, New Jersey
  - Investigational Site Number :8400024, Paramus, New Jersey
  - Investigational Site Number :8400010, New York, New York
  - Investigational Site Number :8400023, Stony Brook, New York
  - Investigational Site Number :8400009, Winston-Salem, North Carolina
  - Investigational Site Number :8400067, Tigard, Oregon
  - Investigational Site Number :8400001, Pittsburgh, Pennsylvania
  - Investigational Site Number :8400073, Austin, Texas
  - Investigational Site Number :8400072, Dallas, Texas
  - Investigational Site Number :8400070, Dallas, Texas
  - Investigational Site Number :8400080, Denton, Texas
  - Investigational Site Number :8400061, Houston, Texas
  - Investigational Site Number :8400068, Houston, Texas
  - Investigational Site Number :8400084, Plano, Texas
  - Investigational Site Number :8400086, The Woodlands, Texas
  - Investigational Site Number :8400078, Waco, Texas
  - Investigational Site Number :8400082, Webster, Texas
  - Investigational Site Number :8400085, Blacksburg, Virginia
  - Investigational Site Number :8400069, Winchester, Virginia
- Argentina (10):
  - Investigational Site Number :0320001, CABA, Buenos Aires
  - Investigational Site Number :0320005, CABA, Buenos Aires
  - Investigational Site Number :0320008, Capital Federal, Buenos Aires
  - Investigational Site Number :0320006, Pergamino, Buenos Aires
  - Investigational Site Number :0320010, Córdoba, Córdoba Province
  - Investigational Site Number :0320002, Rosario, Santa Fe Province
  - Investigational Site Number :0320004, Buenos Aires
  - Investigational Site Number :0320003, La Rioja
  - Investigational Site Number :0320009, Mar del Plata
  - Investigational Site Number :0320007, Salta
- Australia (5):
  - Investigational Site Number :0360004, Macquarie Park, New South Wales
  - Investigational Site Number :0360005, Randwick, New South Wales
  - Investigational Site Number :0360003, Wahroonga, New South Wales
  - Investigational Site Number :0360002, Richmond, Victoria
  - Investigational Site Number :0360001, Nedlands, Western Australia
- Investigational Site Number :0400001, Graz, Austria
- Belgium (4):
  - Investigational Site Number :0560003, Brussels
  - Investigational Site Number :0560004, Charleroi
  - Investigational Site Number :0560001, Leuven
  - Investigational Site Number :0560002, Namur
- Brazil (6):
  - Investigational Site Number :0760005, Porto Alegre, Rio Grande do Sul
  - Investigational Site Number :0760006, Porto Alegre, Rio Grande do Sul
  - Investigational Site Number :0760007, São Paulo, São Paulo
  - Investigational Site Number :0760003, São Paulo, São Paulo
  - Investigational Site Number :0760004, Rio de Janeiro
  - Investigational Site Number :0760008, São Paulo
- Bulgaria (4):
  - Investigational Site Number :1000004, Burgas
  - Investigational Site Number :1000005, Dobrich
  - Investigational Site Number :1000008, Rousse
  - Investigational Site Number :1000001, Sofia
- Canada (5):
  - Investigational Site Number :1240004, Kingston, Ontario
  - Investigational Site Number :1240002, Toronto, Ontario
  - Investigational Site Number :1240007, Greenfield Park, Quebec
  - Investigational Site Number :1240014, Montreal, Quebec
  - Investigational Site Number :1240005, Montreal, Quebec
- Chile (9):
  - Investigational Site Number :1520005, La Serena, Coquimbo Region
  - Investigational Site Number :1520004, Temuco, La Araucanía
  - Investigational Site Number :1520009, Talca, Maule Region
  - Investigational Site Number :1520011, Santaigo, Reg Metropolitana de Santiago
  - Investigational Site Number :1520006, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number :1520002, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number :1520001, Viña del Mar, Región de Valparaíso
  - Investigational Site Number :1520007, Santiago
  - Investigational Site Number :1520003, Santiago
- China (34):
  - Investigational Site Number :1560038, Baoding
  - Investigational Site Number :1560008, Beijing
  - Investigational Site Number :1560035, Beijing
  - Investigational Site Number :1560003, Changchun
  - Investigational Site Number :1560036, Changchun
  - Investigational Site Number :1560013, Chengdu
  - Investigational Site Number :1560019, Chongqing
  - Investigational Site Number :1560031, Dalian
  - Investigational Site Number :1560021, Dalian
  - Investigational Site Number :1560054, Deyang
  - Investigational Site Number :1560043, Fuzhou
  - Investigational Site Number :1560025, Guangzhou
  - Investigational Site Number :1560006, Hangzhou
  - Investigational Site Number :1560007, Hangzhou
  - Investigational Site Number :1560002, Hangzhou
  - Investigational Site Number :1560005, Hangzhou
  - Investigational Site Number :1560011, Harbin
  - Investigational Site Number :1560041, Hefei
  - Investigational Site Number :1560018, Jinan
  - Investigational Site Number :1560046, Jinan
  - Investigational Site Number :1560051, Jining
  - Investigational Site Number :1560017, Linyi
  - Investigational Site Number :1560055, Luoyang
  - Investigational Site Number :1560048, Neijiang
  - Investigational Site Number :1560001, Shanghai
  - Investigational Site Number :1560037, Shaoguan
  - Investigational Site Number :1560028, Tianjin
  - Investigational Site Number :1560033, Wuhan
  - Investigational Site Number :1560024, Wuhan
  - Investigational Site Number :1560045, Xi'an
  - Investigational Site Number :1560044, Xi'an
  - Investigational Site Number :1560027, Xuzhou
  - Investigational Site Number :1560049, Yantai
  - Investigational Site Number :1560022, Zhengzhou
- Czechia (2):
  - Investigational Site Number :2030001, Brno
  - Investigational Site Number :2030002, Prague
- Finland (3):
  - Investigational Site Number :2460001, Helsinki
  - Investigational Site Number :2460002, Tampere
  - Investigational Site Number :2460003, Turku
- France (9):
  - Investigational Site Number :2500009, Nice
  - Investigational Site Number :2500003, Paris
  - Investigational Site Number :2500001, Paris
  - Investigational Site Number :2500006, Poitiers
  - Investigational Site Number :2500007, Saint-Cloud
  - Investigational Site Number :2500002, Saint-Herblain
  - Investigational Site Number :2500010, Strasbourg
  - Investigational Site Number :2500005, Toulouse
  - Investigational Site Number :2500004, Villejuif
- Georgia (7):
  - Investigational Site Number :2680005, Batumi
  - Investigational Site Number :2680006, Kutaisi
  - Investigational Site Number :2680001, Tbilisi
  - Investigational Site Number :2680002, Tbilisi
  - Investigational Site Number :2680004, Tbilisi
  - Investigational Site Number :2680007, Tbilisi
  - Investigational Site Number :2680003, Tbilisi
- Germany (4):
  - Investigational Site Number :2760006, Bottrop
  - Investigational Site Number :2760003, Münster
  - Investigational Site Number :2760007, Oldenburg in Holstein
  - Investigational Site Number :2760001, Ulm
- Hungary (7):
  - Investigational Site Number :3480008, Budapest
  - Investigational Site Number :3480005, Győr
  - Investigational Site Number :3480011, Gyula
  - Investigational Site Number :3480003, Kaposvár
  - Investigational Site Number :3480009, Kecskemét
  - Investigational Site Number :3480010, Miskolc
  - Investigational Site Number :3480001, Nyíregyháza
- Italy (8):
  - Investigational Site Number :3800008, Meldola (FC), Emilia-Romagna
  - Investigational Site Number :3800003, Rozzano, Milano
  - Investigational Site Number :3800007, Monza, Monza E Brianza
  - Investigational Site Number :3800010, Bologna
  - Investigational Site Number :3800004, Milan
  - Investigational Site Number :3800002, Milan
  - Investigational Site Number :3800006, Napoli
  - Investigational Site Number :3800005, Prato
- Japan (20):
  - Investigational Site Number :3920016, Nagoya, Aichi-ken
  - Investigational Site Number :3920007, Nagoya, Aichi-ken
  - Investigational Site Number :3920002, Kashiwa-shi, Chiba
  - Investigational Site Number :3920009, Matsuyama, Ehime
  - Investigational Site Number :3920019, Kurume-shi, Fukuoka
  - Investigational Site Number :3920017, Takasaki-shi, Gunma
  - Investigational Site Number :3920010, Hiroshima, Hiroshima
  - Investigational Site Number :3920001, Sapporo, Hokkaido
  - Investigational Site Number :3920012, Kagoshima, Kagoshima-ken
  - Investigational Site Number :3920014, Yokohama, Kanagawa
  - Investigational Site Number :3920006, Yokohama, Kanagawa
  - Investigational Site Number :3920020, Sendai, Miyagi
  - Investigational Site Number :3920022, Miyazaki, Miyazaki
  - Investigational Site Number :3920008, Osaka, Osaka
  - Investigational Site Number :3920018, Osaka, Osaka
  - Investigational Site Number :3920013, Hidaka-shi, Saitama
  - Investigational Site Number :3920021, Shizuoka, Shizuoka
  - Investigational Site Number :3920003, Koto-ku, Tokyo
  - Investigational Site Number :3920015, Meguro-ku, Tokyo
  - Investigational Site Number :3920005, Shinagawa-ku, Tokyo
- Netherlands (3):
  - Investigational Site Number :5280006, Arnhem
  - Investigational Site Number :5280005, Delft
  - Investigational Site Number :5280001, Maastricht
- Poland (2):
  - Investigational Site Number :6160007, Poznan, Greater Poland Voivodeship
  - Investigational Site Number :6160002, Tomaszów Mazowiecki, Lódzkie
- Portugal (3):
  - Investigational Site Number :6200005, Almada
  - Investigational Site Number :6200001, Lisbon
  - Investigational Site Number :6200002, Porto
- Russia (9):
  - Investigational Site Number :6430007, Arkhangelsk
  - Investigational Site Number :6430004, Krasnogorskiy District
  - Investigational Site Number :6430008, Moscow
  - Investigational Site Number :6430003, Moscow
  - Investigational Site Number :6430005, Moscow
  - Investigational Site Number :6430006, Moscow
  - Investigational Site Number :6430009, Moscow Region
  - Investigational Site Number :6430001, Saint Petersburg
  - Investigational Site Number :6430010, Saint Petersburg
- Singapore (3):
  - Investigational Site Number :7020002, Singapore
  - Investigational Site Number :7020004, Singapore
  - Investigational Site Number :7020001, Singapore
- South Africa (2):
  - Investigational Site Number :7100004, Cape Town
  - Investigational Site Number :7100006, Johannesburg
- South Korea (9):
  - Investigational Site Number :4100006, Goyang-si, Gyeonggi-do
  - Investigational Site Number :4100005, Seongnam-si, Gyeonggi-do
  - Investigational Site Number :4100007, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number :4100004, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number :4100003, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number :4100002, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number :4100001, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number :4100009, Seochogu
  - Investigational Site Number :4100008, Seongnam-si, Gyeonggi-do
- Spain (10):
  - Investigational Site Number :7240011, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number :7240008, Barcelona / Sabadell, Castille and León
  - Investigational Site Number :7240003, Santiago de Compostela, Galicia [Galicia]
  - Investigational Site Number :7240004, Madrid, Madrid, Comunidad de
  - Investigational Site Number :7240006, Madrid / Madrid, Madrid, Comunidad de
  - Investigational Site Number :7240002, Madrid / Madrid, Madrid, Comunidad de
  - Investigational Site Number :7240005, Valencia, Valenciana, Comunidad
  - Investigational Site Number :7240001, Madrid
  - Investigational Site Number :7240007, Málaga
  - Investigational Site Number :7240009, Valencia
- Taiwan (4):
  - Investigational Site Number :1580007, Kaohsiung City
  - Investigational Site Number :1580002, Tainan
  - Investigational Site Number :1580001, Taipei
  - Investigational Site Number :1580003, Taipei
- Turkey (Türkiye) (13):
  - Investigational Site Number :7920006, Adana
  - Investigational Site Number :7920008, Ankara
  - Investigational Site Number :7920009, Ankara
  - Investigational Site Number :7920007, Antalya
  - Investigational Site Number :7920005, Bornova
  - Investigational Site Number :7920013, Diyarbakır
  - Investigational Site Number :7920003, Edirne
  - Investigational Site Number :7920001, Istanbul
  - Investigational Site Number :7920011, Istanbul
  - Investigational Site Number :7920004, Istanbul
  - Investigational Site Number :7920012, Izmir
  - Investigational Site Number :7920010, Kocaeli
  - Investigational Site Number :7920002, Malatya
- Ukraine (5):
  - Investigational Site Number :8040004, Kharkiv
  - Investigational Site Number :8040010, Kharkiv
  - Investigational Site Number :8040001, Kryvyi Rih
  - Investigational Site Number :8040002, Odesa
  - Investigational Site Number :8040007, Vinnytsia
- United Kingdom (3):
  - Investigational Site Number :8260001, Glasgow, Central Bedfordshire
  - Investigational Site Number :8260002, Edinburgh, Edinburgh, City of
  - Investigational Site Number :8260005, Blackburn, Lancashire

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Cortes J, Hurvitz SA, O'Shaughnessy J, Delaloge S, Iwata H, Rugo HS, Neven P, Kanagavel D, Cohen P, Paux G, Cartot-Cotton S, Stefanova-Urena M, Deyme L, Aouni J, Sebastien B, Bardia A. Randomized Phase III Study of Amcenestrant Plus Palbociclib Versus Letrozole Plus Palbociclib in Estrogen Receptor-Positive, Human Epidermal Growth Factor Receptor 2-Negative Advanced Breast Cancer: Primary Results From AMEERA-5. J Clin Oncol. 2024 Aug 1;42(22):2680-2690. doi: 10.1200/JCO.23.02036. Epub 2024 Jun 18. PMID 38889373
- [Derived] Bardia A, Cortes J, Hurvitz SA, Delaloge S, Iwata H, Shao ZM, Kanagavel D, Cohen P, Liu Q, Cartot-Cotton S, Pelekanou V, O'Shaughnessy J. AMEERA-5: a randomized, double-blind phase 3 study of amcenestrant plus palbociclib versus letrozole plus palbociclib for previously untreated ER+/HER2- advanced breast cancer. Ther Adv Med Oncol. 2022 Mar 15;14:17588359221083956. doi: 10.1177/17588359221083956. eCollection 2022. PMID 35309087
- See also: EFC15935 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25234&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 249 active sites in 30 countries. A total of 1277 participants were screened between 14 October 2020 and 11 November 2021, of which 209 were screen failures. Screen failures were mainly due to not meeting selection criteria.
Pre-assignment Details: A total of 1068 participants were randomized, of which 2 participants were randomized but not exposed to study treatment. Randomization was stratified by De-novo metastatic disease (Yes or No); postmenopausal women (Yes or No); visceral metastasis defined by at least 1 liver, lung, brain metastasis, pleural, or peritoneal involvement (Yes or No).
Groups:
- Letrozole + Palbociclib: Participants received letrozole 2.5 milligram (mg) capsule along with amcenestrant-matching placebo once daily, continuously and palbociclib 125 mg orally (PO), once daily (QD) from Day 1 to Day 21 of each 28-day treatment cycle until disease progression, death or study cut-off date, whichever comes first (maximum exposure: 112 weeks).
- Amcenestrant + Palbociclib: Participants received amcenestrant 200 mg tablet along with letrozole-matching placebo once daily, continuously and palbociclib 125 mg PO, QD from Day 1 to Day 21 of each 28-day treatment cycle until disease progression, death, or study cut-off date, whichever comes first (maximum exposure: 109 weeks).
Period: Overall Study
Arm/Group | Letrozole + Palbociclib | Amcenestrant + Palbociclib
Started | 534 | 534
Treated | 533 | 533
Completed | 0 | 0
Not Completed | 534 | 534
Not completed — Adverse Event | 20 | 21
Not completed — Progressive disease | 146 | 168
Not completed — Poor compliance to protocol | 1 | 0
Not completed — Withdrawal by Subject | 19 | 16
Not completed — Data Monitoring Committee recommendation due to negative interim analysis | 309 | 286
Not completed — Study terminated by sponsor | 33 | 35
Not completed — Other: unspecified | 5 | 7
Not completed — Randomized but not treated | 1 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on safety population which included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention, analyzed according to the treatment arm they actually received.
Groups:
- Letrozole + Palbociclib: Participants received letrozole 2.5 mg capsule along with amcenestrant-matching placebo once daily, continuously and palbociclib 125 mg, PO, QD from Day 1 to Day 21 of each 28-day treatment cycle until disease progression, death or study cut-off date, whichever comes first (maximum exposure: 112 weeks).
- Amcenestrant + Palbociclib: Participants received amcenestrant 200 mg tablet along with letrozole-matching placebo once daily, continuously and palbociclib 125 mg PO, QD from Day 1 to Day 21 of each 28-day treatment cycle until disease progression, death or study cut-off date, whichever comes first (maximum exposure: 109 weeks).
- Total: Total of all reporting groups
Arm/Group | Letrozole + Palbociclib | Amcenestrant + Palbociclib | Total
Number analyzed (Participants) | 533 | 533 | 1066
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (12.3) | 57.8 (12.1) | 57.6 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 529 | 524 | 1053
  Male | 4 | 9 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 179 | 175 | 354
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 10 | 10 | 20
  White | 306 | 304 | 610
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 36 | 41 | 77

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time interval (in months) from the date of randomization to the date of first documented tumor progression as per Response Evaluation Criteria in Solid Tumors (RECIST 1.1) assessed by local radiologist or investigator, or death (due to any cause), whichever comes first. Progressive Disease (PD) as per RECIST 1.1: at least a 20 percent (%) increase in sum of diameters of target lesions, unequivocal progression of existing non-target lesions. Analysis was performed by Kaplan-Meier method.
Time Frame: From randomization to the date of first documented tumor progression or death due to any cause or data cut-off date whichever comes first (maximum duration: 81 weeks)
Population: Analysis was performed on the ITT population which included all enrolled participants (i.e., who signed the informed consent form and for whom there was a confirmation of successful allocation of a randomization number by Interactive Response Technology [IRT].
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Letrozole + Palbociclib: Participants received letrozole 2.5 mg capsule along with amcenestrant-matching placebo once daily, continuously and palbociclib 125 mg PO, QD from Day 1 to Day 21 of each 28-day treatment cycle until disease progression, death or study cut-off date, whichever comes first (maximum exposure: 112 weeks).
Arm/Group | Letrozole + Palbociclib | Amcenestrant + Palbociclib
Number analyzed (Participants) | 534 | 534
months | 16.6 [14.1 to NA] — Upper limit of 95% confidence interval (CI) was not estimable due to the smaller number of participants with events. | 14.1 [13.9 to NA] — Upper limit of 95% confidence interval (CI) was not estimable due to the smaller number of participants with events.
Statistical Analysis 1: Comparison: Letrozole + Palbociclib vs Amcenestrant + Palbociclib; A hierarchical testing procedure was used to ensure a strong control of the overall Type I error. Testing was then performed sequentially in order the outcome measures were reported and continued when previous outcome measure was statistically significant at one-sided 2.5% for the primary and the first secondary outcome; Test type: Superiority; p = 0.9304, Stratified Log-Rank test — One-sided p-value based on Stratified log-rank test. Threshold for statistical significance at 0.025 level; Stratified on presence of De-novo metastatic disease, Postmenopausal women and Visceral metastasis according to IRT; Hazard Ratio (HR) = 1.209, 95% CI 2-sided [0.939 to 1.557] — Letrozole + Palbociclib versus Amcenestrant + Palbociclib

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the interval (in months) from the date of randomization to the date of documented death (due to any cause). In the absence of observation of death, survival time was censored to last date the participant was known to be alive or at the cut-off date, whichever comes first. Analysis was performed by Kaplan-Meier method.
Time Frame: From randomization to the death due to any cause or data cut-off date, whichever comes first (maximum duration: 81 weeks)
Population: Analysis was performed on the ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Letrozole + Palbociclib | Amcenestrant + Palbociclib
Number analyzed (Participants) | 534 | 534
months | NA [NA to NA] — Median, upper limit and lower limit of 95% CI were not estimable due to the smaller number of participants with events. | NA [NA to NA] — Median, upper limit and lower limit of 95% CI were not estimable due to the smaller number of participants with events.

3. Secondary Outcome: 12-month Progression-free Survival (PFS) Rate
Description: Percentage of participants who were disease progression-free at Month 12 after randomization were reported in this outcome measure. PFS was defined as the time interval (in months) from the date of randomization to the date of first documented tumor progression as per RECIST 1.1 assessed by local radiologist or investigator, or death (due to any cause), whichever comes first. PD as per RECIST 1.1: at least a 20% increase in sum of diameters of target lesions, unequivocal progression of existing non-target lesions. The PFS rate at Month 12 was estimated using the Kaplan-Meier method and provided an estimation of the percentage of participants who were disease progression-free at Month 12 after randomization.
Time Frame: Month 12
Population: Analysis was performed on the ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Letrozole + Palbociclib | Amcenestrant + Palbociclib
Number analyzed (Participants) | 534 | 534
percentage of participants | 68.2 [61.2 to 74.2] | 65.5 [59.1 to 71.1]

4. Secondary Outcome: Percentage of Participants With Objective Response
Description: Objective response was defined as percentage of participants having a partial response (PR) or complete response (CR) according to the RECIST version 1.1 assessed by investigator. As per RECIST 1.1, CR was defined as disappearance of all target and non-target lesions and normalization of tumor marker level. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<) 10 millimeters (mm). PR was defined as at least a 30%decrease in the sum of diameters of target lesions, taking as reference the Baseline sum diameters.
Time Frame: From randomization to the date of first documented tumor progression, death due to any cause or data cut-off date whichever comes first (maximum duration: 81 weeks)
Population: Analysis was performed on the ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Letrozole + Palbociclib | Amcenestrant + Palbociclib
Number analyzed (Participants) | 534 | 534
percentage of participants | 42.3 [38.1 to 46.6] | 32.2 [28.3 to 36.4]

5. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as time (in months) from first documented evidence of CR or PR until disease progression determined by investigator as per RECIST 1.1, or start of any anti-cancer therapy, or death from any cause, whichever occurs first. For participants with ongoing response at the time of the analysis, DOR was censored at the date of the last valid disease assessment not showing documented progression performed before the initiation of a new anticancer treatment (if any). As per RECIST 1.1, CR was defined as disappearance of all target and non-target lesions and normalization of tumor marker level. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the Baseline sum diameters. PD: at least 20% increase in sum of diameters of target lesions, unequivocal progression of existing non-target lesions. Analysis was performed by Kaplan-Meier method.
Time Frame: From the date of first response of CR or PR until disease progression or death, or start of any anti-cancer therapy or data cut-off date, whichever comes first (maximum duration: 81 weeks)
Population: Analysis was performed on a subset of participants who had objective response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Letrozole + Palbociclib | Amcenestrant + Palbociclib
Number analyzed (Participants) | 226 | 172
months | 14.0 [11.1 to NA] — Upper limit of 95% CI was not estimable due to small number of progression events or death. | NA [11.4 to NA] — Median and upper limit of 95% CI was not estimable due to the small number of progression events or death.

6. Secondary Outcome: Percentage of Participants With Clinical Benefit
Description: Clinical Benefit was defined as the percentage of participants having a confirmed CR, PR, or stable disease (SD) for at least 24 weeks determined by investigator as per RECIST 1.1, from date of randomization until disease progression, or death, or data cut-off date, or initiation of post treatment anti-cancer therapy, whichever occurs first. As per RECIST 1.1; CR was defined as disappearance of all target, non-target lesions & normalization of tumor marker level. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: at least a 30% decrease in sum of diameters of target lesions, taking as reference Baseline sum diameters. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference smallest sum diameters. PD: at least 20% increase in sum of diameters of target lesions, unequivocal progression of existing non-target lesions.
Time Frame: From randomization until disease progression, or death, or data cut-off date, whichever comes first (maximum duration: 81 weeks)
Population: Analysis was performed on the ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Letrozole + Palbociclib | Amcenestrant + Palbociclib
Number analyzed (Participants) | 534 | 534
percentage of participants | 82.4 [78.9 to 85.5] | 76.0 [72.2 to 79.6]

7. Secondary Outcome: Progression-free Survival on Next Line of Therapy (PFS2)
Description: PFS2 was defined as the time interval (in months) from the date of randomization to the date of first documentation of PD on the next systemic anti-cancer therapy according to investigator, or death due to any cause in the absence of documented PD on the next systemic anti-cancer therapy, whichever occurs first. PD was defined as at least 20% increase in sum of diameters of target lesions, unequivocal progression of existing non-target lesions. Analysis was performed by Kaplan-Meier method.
Time Frame: From randomization to date first documented disease progression on the next systemic anti-cancer therapy, or death due to any cause, or data cut-off date, whichever comes first (maximum duration: 81 weeks)
Population: Analysis was performed on the ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Letrozole + Palbociclib | Amcenestrant + Palbociclib
Number analyzed (Participants) | 534 | 534
months | NA [NA to NA] — Median, upper and lower limit of 95% CI was not estimable due to the smaller number of participants with events. | NA [NA to NA] — Median, upper and lower limit of 95% CI was not estimable due to the smaller number of participants with events.

8. Secondary Outcome: Pharmacokinetics: Plasma Concentrations of Amcenestrant
Description: Amcenestrant plasma concentrations at specified time points were reported. Data for this outcome measure was not planned to be collected and analyzed for Letrozole+Palbociclib arm as pre-specified in protocol.
Time Frame: Cycle 1 Day 1: 3 hours (hr) post-dose, Cycle 1 Day 15: pre-dose, Cycle 2 Day 1: pre-dose, 3 hr post-dose, Cycle 2 Day 15: pre-dose, Cycle 3 Day 1: pre-dose, Cycle 4 Day 1: pre-dose, Cycle 7 Day 1: pre-dose, Cycle 10 Day 1: pre-dose
Population: Analysis was performed on the Pharmacokinetic-evaluable (amcenestrant) population that included all participants who took at least 1 dose of study intervention, and with at least one evaluable plasma concentration of amcenestrant post-treatment. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure and 'Number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Arm/Group | Amcenestrant + Palbociclib
Number analyzed (Participants) | 531
nanograms per milliliter
  Cycle 1 Day 1: 3 hr post-dose: number analyzed (Participants) | 473
  Cycle 1 Day 1: 3 hr post-dose | 2890.0 (1783.8)
  Cycle 1 Day 15: pre-dose: number analyzed (Participants) | 283
  Cycle 1 Day 15: pre-dose | 399.5 (575.0)
  Cycle 2 Day 1: pre-dose: number analyzed (Participants) | 255
  Cycle 2 Day 1: pre-dose | 387.5 (685.6)
  Cycle 2 Day 1: 3 hr post-dose: number analyzed (Participants) | 441
  Cycle 2 Day 1: 3 hr post-dose | 2729.3 (1604.4)
  Cycle 2 Day 15: pre-dose: number analyzed (Participants) | 253
  Cycle 2 Day 15: pre-dose | 361.3 (572.8)
  Cycle 3 Day 1: pre-dose: number analyzed (Participants) | 215
  Cycle 3 Day 1: pre-dose | 303.4 (315.7)
  Cycle 4 Day 1: pre-dose: number analyzed (Participants) | 169
  Cycle 4 Day 1: pre-dose | 349.3 (385.3)
  Cycle 7 Day 1: pre-dose: number analyzed (Participants) | 162
  Cycle 7 Day 1: pre-dose | 337.5 (432.9)
  Cycle 10 Day 1: pre-dose: number analyzed (Participants) | 118
  Cycle 10 Day 1: pre-dose | 310.9 (253.3)

9. Secondary Outcome: Pharmacokinetics: Plasma Concentrations of Palbociclib
Description: Palbociclib plasma concentrations at specified time points were reported.
Time Frame: Cycle 1 Day 1: 3 hr post-dose, Cycle 1 Day 15: pre-dose, Cycle 2 Day 1: pre-dose, 3 hr post-dose, Cycle 2 Day 15: pre-dose, Cycle 3 Day 1: pre-dose, Cycle 4 Day 1: pre-dose, Cycle 7 Day 1: pre-dose, Cycle 10 Day 1: pre-dose
Population: Analysis was performed on the Pharmacokinetic-evaluable (palbociclib) population that included all participants who took at least 1 dose of study intervention, and with at least one evaluable plasma concentration of palbociclib post-treatment. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Arm/Group | Letrozole + Palbociclib | Amcenestrant + Palbociclib
Number analyzed (Participants) | 532 | 532
nanograms per milliliter
  Cycle 1 Day 1: 3 hr post-dose: number analyzed (Participants) | 479 | 472
  Cycle 1 Day 1: 3 hr post-dose | 36.265 (31.110) | 37.780 (31.005)
  Cycle 1 Day 15: pre-dose: number analyzed (Participants) | 264 | 274
  Cycle 1 Day 15: pre-dose | 82.541 (38.671) | 45.903 (20.086)
  Cycle 2 Day 1: pre-dose: number analyzed (Participants) | 201 | 227
  Cycle 2 Day 1: pre-dose | 3.409 (8.498) | 2.159 (7.368)
  Cycle 2 Day 1: 3 hr post-dose: number analyzed (Participants) | 316 | 385
  Cycle 2 Day 1: 3 hr post-dose | 30.234 (26.967) | 27.144 (24.667)
  Cycle 2 Day 15: pre-dose: number analyzed (Participants) | 237 | 247
  Cycle 2 Day 15: pre-dose | 72.176 (35.210) | 42.882 (18.081)
  Cycle 3 Day 1: pre-dose: number analyzed (Participants) | 183 | 192
  Cycle 3 Day 1: pre-dose | 4.301 (11.796) | 1.615 (4.283)
  Cycle 4 Day 1: pre-dose: number analyzed (Participants) | 131 | 150
  Cycle 4 Day 1: pre-dose | 4.767 (17.787) | 1.390 (3.052)
  Cycle 7 Day 1: pre-dose: number analyzed (Participants) | 143 | 142
  Cycle 7 Day 1: pre-dose | 2.716 (2.058) | 1.461 (1.722)
  Cycle 10 Day 1: pre-dose: number analyzed (Participants) | 97 | 102
  Cycle 10 Day 1: pre-dose | 3.793 (7.675) | 1.489 (1.155)

10. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC-QLQ-C30) Domain Scores
Description: EORTC-QLQ-C30: cancer-specific instrument with 30 questions for evaluation of new chemotherapy & assessment of participant reported outcome. These include 5 functional scales, 9 symptom scales, & Global Health Status/quality of life scale (GHS/QoL). All 14 items/domains were scored on scale of 1 (not at all) to 4 (very much) & GHS/QoL, scored on scale of 1 (very poor) to 7 (excellent). All scales are transformed from raw scores to linear scales ranging 0 to 100. Higher score for functional & GHS/QoL=higher level of functioning, & higher score for symptoms scales=higher symptom burden. Least Square (LS) mean and Standard Error (SE) were derived from MMRM model with change from Baseline values as response variable, treatment, time, treatment-by-time interaction, Baseline value and stratifications factors as fixed effect. Average of LS mean change from Baseline values of overall treatment (i.e., each cycle [Cycle 1 up to Cycle 21]) for each domain was reported in this outcome measure.
Time Frame: Baseline, overall treatment duration (Cycle 1 up to Cycle 21 [i.e., 81 weeks])
Population: Analysis was performed on safety population. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Letrozole + Palbociclib | Amcenestrant + Palbociclib
Number analyzed (Participants) | 533 | 533
score on a scale
  GHS/QoL: number analyzed (Participants) | 491 | 485
  GHS/QoL | 2.8 (0.6) | 3.1 (0.6)
  Physical functioning: number analyzed (Participants) | 488 | 484
  Physical functioning | 2.3 (0.5) | 2.6 (0.6)
  Role functioning: number analyzed (Participants) | 490 | 482
  Role functioning | 1.8 (0.7) | 2.0 (0.7)
  Emotional functioning: number analyzed (Participants) | 490 | 484
  Emotional functioning | 4.2 (0.6) | 4.1 (0.7)
  Cognitive functioning: number analyzed (Participants) | 491 | 485
  Cognitive functioning | -0.8 (0.6) | -1.2 (0.6)
  Social functioning: number analyzed (Participants) | 489 | 485
  Social functioning | 2.2 (0.7) | 4.4 (0.8)
  Fatigue: number analyzed (Participants) | 490 | 484
  Fatigue | -1.6 (0.7) | -2.0 (0.7)
  Nausea and vomiting: number analyzed (Participants) | 485 | 478
  Nausea and vomiting | -1.3 (0.4) | -0.6 (0.4)
  Pain: number analyzed (Participants) | 491 | 485
  Pain | -5.8 (0.7) | -6.8 (0.7)
  Dyspnea: number analyzed (Participants) | 488 | 480
  Dyspnea | -1.1 (0.7) | -0.7 (0.7)
  Insomnia: number analyzed (Participants) | 490 | 483
  Insomnia | -2.9 (0.9) | -3.9 (0.9)
  Appetite loss: number analyzed (Participants) | 485 | 478
  Appetite loss | -3.0 (0.7) | -2.7 (0.7)
  Constipation: number analyzed (Participants) | 486 | 477
  Constipation | 0.1 (0.8) | 0.0 (0.9)
  Diarrhea: number analyzed (Participants) | 490 | 480
  Diarrhea | -0.4 (0.4) | 0.4 (0.4)
  Financial difficulties: number analyzed (Participants) | 488 | 485
  Financial difficulties | -5.1 (0.8) | -4.0 (0.8)

11. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Breast Cancer Specific Module (EORTC-QLQ-BR23) Domain Scores
Description: QLQ-BR23: disease-specific Health-related QOL assesses breast cancer impact & side effects of treatment. EORTCQLQ- BR23 contains 23 items: multi-item scales & single-item measures. 4 functional scales (body image, sexual functioning, sexual enjoyment, future perspective) & 4 scales related to symptoms of disease or treatment (arm symptoms, breast symptoms, systemic therapy side effects, & upset by hair loss). All items scored 1 (not at all) to 4 (very much). Scores of all scales transformed from raw scores to linear scales ranging 0-100. Higher score for functional scales=better outcome; higher score for symptoms scales=higher symptom burden. LS mean & SE were derived from MMRM model with change from Baseline values as response variable, treatment, time, treatment-by-time interaction, Baseline value & stratifications factors as fixed effect. Average of LS mean change from Baseline values of overall treatment (i.e., each cycle [Cycle 1 up to Cycle 21]) for each domain was reported.
Time Frame: Baseline, overall treatment duration (Cycle 1 up to Cycle 21 [i.e., 81 weeks])
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Letrozole + Palbociclib | Amcenestrant + Palbociclib
Number analyzed (Participants) | 533 | 533
score on a scale
  Body image: number analyzed (Participants) | 463 | 464
  Body image | 1.3 (0.7) | 1.1 (0.7)
  Sexual functioning: number analyzed (Participants) | 451 | 450
  Sexual functioning | -1.4 (0.6) | -1.5 (0.6)
  Sexual enjoyment: number analyzed (Participants) | 101 | 98
  Sexual enjoyment | -10.4 (1.9) | -8.7 (1.9)
  Future perspective: number analyzed (Participants) | 467 | 465
  Future perspective | 11.6 (1.0) | 10.8 (1.0)
  Systemic therapy side effects: number analyzed (Participants) | 466 | 466
  Systemic therapy side effects | 4.9 (0.5) | 3.7 (0.5)
  Breast symptoms: number analyzed (Participants) | 466 | 465
  Breast symptoms | -7.6 (0.5) | -7.0 (0.5)
  Arm symptoms: number analyzed (Participants) | 466 | 466
  Arm symptoms | -1.9 (0.6) | -1.8 (0.6)
  Upset by hair loss: number analyzed (Participants) | 89 | 75
  Upset by hair loss | -2.7 (2.2) | -0.2 (2.5)

12. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Breast Cancer Specific Module (EORTC QLQ-BR45) Domain Scores
Description: EORTC QLQ-BR45: comprised of all 23 items from the QLQ-BR23 plus an additional 22 items assessing endocrine therapy symptoms (10 items), endocrine sexual symptoms (4 items), breast satisfaction (2 items), and skin mucosis symptoms (6 items). All items scored 1 (not at all) to 4 (very much). Scores of all scales transformed from raw scores to linear scales ranging 0 to 100. Higher score for functional scales = better outcome; higher score for symptoms scales = higher symptom burden. LS mean and SE are derived from Mixed Model Repeated Measures (MMRM) model with change from Baseline values as response variable, treatment, time, treatment-by-time interaction, Baseline value and stratifications factors as fixed effect. Average of LS mean change from Baseline values of overall treatment (i.e., each cycle [Cycle 1 up to Cycle 21]) for each domain (endocrine therapy symptoms, endocrine sexual symptoms, breast satisfaction and skin mucosis symptoms) was reported.
Time Frame: Baseline, overall treatment duration (Cycle 1 up to Cycle 21 [i.e., 81 weeks])
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Letrozole + Palbociclib | Amcenestrant + Palbociclib
Number analyzed (Participants) | 533 | 533
score on a scale
  Breast Satisfaction: number analyzed (Participants) | 378 | 369
  Breast Satisfaction | -1.7 (1.2) | 1.0 (1.3)
  Endocrine Sexual Symptoms: number analyzed (Participants) | 428 | 419
  Endocrine Sexual Symptoms | 4.8 (0.8) | 2.3 (0.8)
  Endocrine Therapy Symptoms: number analyzed (Participants) | 437 | 434
  Endocrine Therapy Symptoms | 1.5 (0.6) | 1.2 (0.6)
  Skin Mucosis Symptoms: number analyzed (Participants) | 438 | 434
  Skin Mucosis Symptoms | 3.5 (0.5) | 2.5 (0.5)

13. Secondary Outcome: Change From Baseline in European Quality of Life Working Group Health Status Measure 5 Dimensions (5D), 5 Levels (5L) (EQ-5D-5L) Score: Visual Analog Scale (VAS) Score
Description: EQ-5D-5L is a standardized measure of health status, provides a simple, generic measure of health for clinical and economic appraisal, and consists of 2 sections: the EQ-5D-5L health state utility index (descriptive system) and the EQ-5D-5L VAS. The Visual Analogue Scale is designed to rate the participant's current health state on a scale from 0 to 100, where 0 represents the worst imaginable health state and 100 represents the best imaginable health state. LS mean and SE are derived from MMRM model with change from Baseline values as response variable, treatment, time, treatment-by-time interaction, Baseline value and stratifications factors as fixed effect. Average of LS mean change from Baseline values of overall treatment (i.e., each cycle [Cycle 1 up to Cycle 21]) for VAS was reported in this outcome measure.
Time Frame: Baseline, overall treatment duration (Cycle 1 up to Cycle 21 [i.e., 81 weeks])
Population: Analysis was performed on safety population. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Letrozole + Palbociclib: Participants received letrozole 2.5 mg capsule along with amcenestrant-matching placebo once daily, continuously and palbociclib 125 mg PO, QD from Day 1 to Day 21 of each 28-day treatment cycle and were followed until disease progression, death or study cut-off date, whichever comes first (maximum exposure duration: 112 weeks).
Arm/Group | Letrozole + Palbociclib | Amcenestrant + Palbociclib
Number analyzed (Participants) | 492 | 489
score on a scale | 3.2 (0.5) | 3.8 (0.5)

14. Secondary Outcome: Change From Baseline in European Quality of Life Working Group Health Status Measure 5 Dimensions (5D), 5 Levels (5L) (EQ-5D-5L) Score: Health Utility Index Value Score
Description: EQ-5D-5L: consists of 2 sections: EQ-5D-5L health state utility index (descriptive system) & VAS. The EQ-5D descriptive system consists of 5 dimensions: mobility, self-care, usual activities, pain/discomfort & anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, & extreme problems. Response options are measured with 5-point Likert scale (for 5L version). The EQ-5D-5L responses are converted into single index utility score between 0 to 1, where higher score indicates better health state & lower score indicate worse health state. LS mean and SE were derived from MMRM model with change from Baseline values as response variable, treatment, time, treatment-by-time interaction, Baseline value and stratifications factors as fixed effect. Average of LS mean change from Baseline values overall treatment (i.e., each cycle [Cycle 1 up to Cycle 21]) for health utility index value score was reported in this outcome measure.
Time Frame: Baseline, overall treatment duration (Cycle 1 up to Cycle 21 [i.e., 81 weeks])
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Letrozole + Palbociclib | Amcenestrant + Palbociclib
Number analyzed (Participants) | 492 | 489
score on a scale | 0.0 (0.0) | 0.0 (0.0)

15. Secondary Outcome: Time to First Chemotherapy
Description: Time to chemotherapy was defined as the time interval (in months) from the date of randomization to the start date of the first chemotherapy after disease progression.
Time Frame: From randomization to the start date of the first chemotherapy (maximum duration: 81 weeks)
Population: Analysis was performed on the ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Letrozole + Palbociclib | Amcenestrant + Palbociclib
Number analyzed (Participants) | 534 | 534
months | NA [NA to NA] — Median, upper limit and lower limit of 95% CI was not estimable due to lower number of participants with events. | NA [NA to NA] — Median, upper limit and lower limit of 95% CI was not estimable due to lower number of participants with events.

16. Secondary Outcome: Number of Participants With Hematological Abnormalities During the Treatment Period
Description: Hematological parameters assessed were anemia, lymphocyte count decreased, neutrophil count decreased, white blood cell decreased, platelet count decreased. Parameters were assessed as per the National Cancer Institute Common Terminology Criteria for Adverse Experience version 5.0 (NCI-CTCAE v 5.0), where Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Potentially Life Threatening. Grade refers to the severity of the AEs. Treatment period was defined as the time from the first dose of study treatments up to 30 days after last dose of study treatment.
Time Frame: From first dose of study treatment up to 30 days after last dose of study treatment (maximum duration: 112 weeks)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Letrozole + Palbociclib | Amcenestrant + Palbociclib
Number analyzed (Participants) | 533 | 533
Participants
  Anemia: Grade 1: number analyzed (Participants) | 533 | 532
  Anemia: Grade 1 | 309 | 302
  Anemia: Grade 2: number analyzed (Participants) | 533 | 532
  Anemia: Grade 2 | 108 | 78
  Anemia: Grade 3: number analyzed (Participants) | 533 | 532
  Anemia: Grade 3 | 22 | 17
  Anemia: Grade 4: number analyzed (Participants) | 533 | 532
  Anemia: Grade 4 | 0 | 0
  Lymphocyte count decreased: Grade 1: number analyzed (Participants) | 533 | 532
  Lymphocyte count decreased: Grade 1 | 98 | 101
  Lymphocyte count decreased: Grade 2: number analyzed (Participants) | 533 | 532
  Lymphocyte count decreased: Grade 2 | 138 | 124
  Lymphocyte count decreased: Grade 3: number analyzed (Participants) | 533 | 532
  Lymphocyte count decreased: Grade 3 | 46 | 48
  Lymphocyte count decreased: Grade 4: number analyzed (Participants) | 533 | 532
  Lymphocyte count decreased: Grade 4 | 23 | 22
  Neutrophil count decreased: Grade 1: number analyzed (Participants) | 533 | 532
  Neutrophil count decreased: Grade 1 | 22 | 45
  Neutrophil count decreased: Grade 2: number analyzed (Participants) | 533 | 532
  Neutrophil count decreased: Grade 2 | 150 | 217
  Neutrophil count decreased: Grade 3: number analyzed (Participants) | 533 | 532
  Neutrophil count decreased: Grade 3 | 277 | 199
  Neutrophil count decreased: Grade 4: number analyzed (Participants) | 533 | 532
  Neutrophil count decreased: Grade 4 | 70 | 21
  White blood cell decreased: Grade 1: number analyzed (Participants) | 532 | 531
  White blood cell decreased: Grade 1 | 81 | 146
  White blood cell decreased: Grade 2: number analyzed (Participants) | 532 | 531
  White blood cell decreased: Grade 2 | 279 | 267
  White blood cell decreased: Grade 3: number analyzed (Participants) | 532 | 531
  White blood cell decreased: Grade 3 | 163 | 95
  White blood cell decreased: Grade 4: number analyzed (Participants) | 532 | 531
  White blood cell decreased: Grade 4 | 7 | 3
  Platelet count decreased: Grade 1: number analyzed (Participants) | 533 | 532
  Platelet count decreased: Grade 1 | 285 | 220
  Platelet count decreased: Grade 2: number analyzed (Participants) | 533 | 532
  Platelet count decreased: Grade 2 | 30 | 12
  Platelet count decreased: Grade 3: number analyzed (Participants) | 533 | 532
  Platelet count decreased: Grade 3 | 18 | 8
  Platelet count decreased: Grade 4: number analyzed (Participants) | 533 | 532
  Platelet count decreased: Grade 4 | 8 | 10

17. Secondary Outcome: Number of Participants With Liver Function Abnormalities of Grade 3 and 4 During the Treatment Period
Description: Liver Function parameters assessed were aspartate aminotransferase increased, alanine aminotransferase increased, alkaline phosphatase increased, total bilirubin increased, gamma-glutamyl transferase increased. Parameters were assessed as per the NCI-CTCAE v 5.0, where Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Potentially Life Threatening. Grade refers to the severity of the AEs. Treatment period was defined as the time from the first dose of study treatments up to 30 days after last dose of study treatment. Participants with Grade 3 and 4 liver function abnormalities were reported in this outcome measure.
Time Frame: From first dose of study treatment up to 30 days after last dose of study treatment (maximum duration: 112 weeks)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Letrozole + Palbociclib | Amcenestrant + Palbociclib
Number analyzed (Participants) | 533 | 533
Participants
  Aspartate aminotransferase increased: Grade 3: number analyzed (Participants) | 533 | 532
  Aspartate aminotransferase increased: Grade 3 | 9 | 23
  Aspartate aminotransferase increased: Grade 4: number analyzed (Participants) | 533 | 532
  Aspartate aminotransferase increased: Grade 4 | 0 | 1
  Alanine aminotransferase increased: Grade 3: number analyzed (Participants) | 533 | 532
  Alanine aminotransferase increased: Grade 3 | 12 | 32
  Alanine aminotransferase increased: Grade 4: number analyzed (Participants) | 533 | 532
  Alanine aminotransferase increased: Grade 4 | 1 | 3
  Alkaline phosphatase increased: Grade 3: number analyzed (Participants) | 532 | 532
  Alkaline phosphatase increased: Grade 3 | 3 | 1
  Alkaline phosphatase increased: Grade 4: number analyzed (Participants) | 532 | 532
  Alkaline phosphatase increased: Grade 4 | 0 | 0
  Total bilirubin increased: Grade 3: number analyzed (Participants) | 533 | 532
  Total bilirubin increased: Grade 3 | 3 | 5
  Total bilirubin increased: Grade 4: number analyzed (Participants) | 533 | 532
  Total bilirubin increased: Grade 4 | 0 | 0
  Gamma-GT increased: Grade 3: number analyzed (Participants) | 533 | 532
  Gamma-GT increased: Grade 3 | 9 | 20
  Gamma-GT increased: Grade 4: number analyzed (Participants) | 533 | 532
  Gamma-GT increased: Grade 4 | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse Events (AE) data was collected from Baseline up to 30 days after last dose of study treatment (maximum exposure: 112 weeks), deaths were collected from Baseline up to the end of study (26 May 2023)
Description: Reported SAEs and NSAEs were assessed for safety population. All-Cause Mortality data collected during study was assessed for all randomized participants. Disease progression related death were not reported as AE.
Arm/Group | Letrozole + Palbociclib | Amcenestrant + Palbociclib
All-Cause Mortality (participants affected / at risk) | 41/534 | 45/534
Serious Adverse Events (participants affected / at risk) | 68/533 | 77/533
Other Adverse Events (participants affected / at risk) | 448/533 | 412/533
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Letrozole + Palbociclib (N=533) | Amcenestrant + Palbociclib (N=533)
Appendicitis (Infections and infestations) | 2 (2) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 8 (8) | 4 (4)
Covid-19 Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Device Related Infection (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Focal Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Herpes Zoster (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Paracancerous Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 3 (3) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1)
Adenocarcinoma Of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Diffuse Large B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gallbladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases To Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 4 (5) | 1 (1)
Anaemia Of Malignant Disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Schizophrenia (Psychiatric disorders) | 0 (0) | 1 (1)
Cerebral Infarction (Nervous system disorders) | 2 (2) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 1 (1)
Ischaemic Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Psychomotor Hyperactivity (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 3 (3) | 0 (0)
Acute Left Ventricular Failure (Cardiac disorders) | 0 (0) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1) | 2 (2)
Atrioventricular Block Complete (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Failure (Cardiac disorders) | 2 (2) | 0 (0)
Heart Valve Incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 2 (2) | 3 (3)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Vena Cava Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Asthma-Chronic Obstructive Pulmonary Disease Overlap Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 7 (7)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Abdominal Distension (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Pain Lower (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 2 (2) | 1 (1)
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis Acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1)
Bile Duct Stone (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic Failure (Hepatobiliary disorders) | 1 (1) | 2 (2)
Hepatic Function Abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatorenal Failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 1 (1)
Axillary Mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Spinal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Pyelocaliectasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Ovarian Cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 1 (1)
Disease Progression (General disorders) | 4 (4) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
General Physical Health Deterioration (General disorders) | 0 (0) | 1 (2)
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 1 (1)
Oedema Peripheral (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 3 (4)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 2 (2)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 2 (2)
Blood Follicle Stimulating Hormone Decreased (Investigations) | 0 (0) | 1 (1)
Alcohol Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal Procedural Complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal Stoma Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural Pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Letrozole + Palbociclib (N=533) | Amcenestrant + Palbociclib (N=533)
Covid-19 (Infections and infestations) | 53 (53) | 60 (60)
Urinary Tract Infection (Infections and infestations) | 36 (49) | 38 (62)
Neutropenia (Blood and lymphatic system disorders) | 201 (538) | 113 (231)
Decreased Appetite (Metabolism and nutrition disorders) | 44 (51) | 39 (43)
Insomnia (Psychiatric disorders) | 39 (40) | 40 (46)
Dizziness (Nervous system disorders) | 34 (41) | 28 (34)
Headache (Nervous system disorders) | 65 (79) | 56 (73)
Hot Flush (Vascular disorders) | 82 (86) | 87 (90)
Hypertension (Vascular disorders) | 20 (27) | 31 (42)
Cough (Respiratory, thoracic and mediastinal disorders) | 30 (32) | 30 (34)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 32 (35) | 32 (36)
Abdominal Pain Upper (Gastrointestinal disorders) | 28 (31) | 24 (24)
Constipation (Gastrointestinal disorders) | 68 (84) | 70 (76)
Diarrhoea (Gastrointestinal disorders) | 82 (115) | 62 (74)
Nausea (Gastrointestinal disorders) | 92 (112) | 84 (102)
Stomatitis (Gastrointestinal disorders) | 93 (131) | 64 (88)
Vomiting (Gastrointestinal disorders) | 54 (64) | 39 (51)
Alopecia (Skin and subcutaneous tissue disorders) | 72 (72) | 44 (45)
Arthralgia (Musculoskeletal and connective tissue disorders) | 102 (128) | 110 (136)
Back Pain (Musculoskeletal and connective tissue disorders) | 50 (60) | 45 (50)
Myalgia (Musculoskeletal and connective tissue disorders) | 29 (34) | 27 (30)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 22 (24) | 45 (52)
Asthenia (General disorders) | 46 (57) | 45 (55)
Fatigue (General disorders) | 100 (107) | 93 (107)
Alanine Aminotransferase Increased (Investigations) | 18 (20) | 39 (44)
Neutrophil Count Decreased (Investigations) | 114 (252) | 67 (118)
White Blood Cell Count Decreased (Investigations) | 33 (72) | 17 (20)

LIMITATIONS AND CAVEATS:
The study was terminated based on the review by an independent data monitoring committee of the prespecified interim analysis of the Phase 3 AMEERA-5 efficacy data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2021-09-02): https://cdn.clinicaltrials.gov/large-docs/66/NCT04478266/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-11): https://cdn.clinicaltrials.gov/large-docs/66/NCT04478266/SAP_001.pdf